CLINICAL TRIAL: NCT06042530
Title: Cognitive Impairment and Fatigue After Mild to Moderate COVID-19 - Relation to Biomarkers and Neuronal Network Functions
Brief Title: Cognitive Impairment and Fatigue After Mild to Moderate COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other); Karolinska University Hospital (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Marika Moller, Associate Professor, Danderyd Hospital
Other Study IDs: 2021-03907_Cognition COVID-19
Record Dates: First submitted 2023-09-07; First posted 2023-09-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Post COVID-19 Condition; Cognitive Impairment; Fatigue, Mental
Keywords: cognition; fatigue; COVID-19; neuropsychology; biomarkers; vision; imaging
MeSH Terms: conditions — Cognitive Dysfunction; Mental Fatigue; Fatigue; COVID-19 | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Astrocyte-derived EV, and Hmbg1. Exploratory targeted analyses using panels of cytokines & chemokines and neuroinflammation will also be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID condition: Patients experiencing persisting cognitive dysfunction and fatigue after a SARS-CoV-2 infection, three months or more after the infections
  Interventions: Diagnostic Test: Neuropsychological investigation; Diagnostic Test: Optometric investigation; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Immunological biomarkers
- Non-symptomatic controls: Persons experiencing no symptoms after the SARS-CoV-2 infection or have not been subject for at SARS-CoV-2 infection
  Interventions: Diagnostic Test: Neuropsychological investigation; Diagnostic Test: Optometric investigation; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Immunological biomarkers

INTERVENTIONS:
Diagnostic Test: Neuropsychological investigation — Comprehensive neuropsychological test battery covering logical reasoning, different attention functions, executive functions, visuospatial functions, different memory functions, psychomotor speed, motor functions, and smell identification
Diagnostic Test: Optometric investigation — Extended vision examination including symptom assessment, visual acuity, visual field (confrontation), eye movements, eye teaming and clinical assessment of hypersensitivity to visual stimuli.
Diagnostic Test: Magnetic Resonance Imaging — The MRI sequence protocol includes resting state fMRI before and after the participants do an established 20 min long reaction time measurement paradigm (E-prime). During the paradigm a pseudo-continious arterial spin labeling sequence (pCASL) is acquired for continuous measurement of brain perfusion. Following the functional sequences the imaging protocol also includes a high resolution 3D T1weighted sequence Magnetization Prepared Rapid Gradient Echo (MPRAGE) for brain structure, a high resolution 3D T2-weighted sequence Fluid-Attenuated Inversion Recovery (FLAIR) for pathology and a 3D susceptibility weighted image (SWI) for microvascular abnormalities.
Diagnostic Test: Immunological biomarkers — Venous blood samples (10-20 ml) are taken from the elbow crease. They are drawn in the morning, and the participants are asked to fast for 12 hours prior to sampling. They are also asked to avoid physical activity prior to blood sampling. The samples are drawn into citrated tubes.

SUMMARY:
The primary aim of the project is to map fatigue, cognitive and visual dysfunctions and possible underlying pathophysiological mechanisms in persons with long-term symptoms after a mild to moderate COVID-19 infection. Secondary goals are to study whether covarying factors such as depression and sleep disorders contribute to the results.

DETAILED DESCRIPTION:
The primary aim of the project is to map neuropsychological and visual dysfunctions and possible underlying pathophysiological mechanisms in patients suffering from Post-COVID condition (PCC) after a mild to moderate COVID-19 infection. Secondary goals are to study whether covarying factors such as depression and sleep disorders contribute to the results.

The main objectives are:

1. Which cognitive problems (self-reported and test results/performance based?) are typical in patients with post-COVID syndrome compared to non-symptomatic controls?
2. Which pre-existing factors affect cognitive functions and fatigue after a mild to moderate COVID-19 infection?
3. Is there a relationship between self-perceived symptoms, cognitive and visual test results, optical coherence tomography (OCT) examination, imaging results, and biomarkers in patients who have undergone mild COVID-19 infection and does this differ compared to non-symptomatic controls?
4. How are fatigue, cognitive fatigability and vision-related disorders related to neuronal correlates and changes in the retina examined with OCT and biomarkers (astocyte-derived extracellular vesicles (High Mobility Group Box 1 (Hmbg1) and S100B) and inflammatory markers) in patients who have remaining symptoms after a mild COVID-19 infection and do the results differ from what can be seen in non-symptomatic controls?
5. Are specific cognitive dysfunctions and fatigue/cognitive fatigability correlated with astocyte-derived extracellular vesicles in patients who have remaining symptoms after a mild COVID-19 infection?
6. How do symptoms evolve over one and two years?

STUDY DESIGN The study is a controlled longitudinal cohort study that includes cross-sectional sub-studies of imaging and biomarkers.

STUDY SETTING Outpatient rehabilitation clinic at the Department of Rehabilitation Medicine at Danderyd University Hospital and Karolinska University Hospital, both located in Stockholm, Sweden. At the Cognitive post-COVID clinic at Danderyd University Hospital, patients with long-term cognitive problems and fatigue are investigated after a mild to moderat (not ICU treated) COVID-19 infection. Clinical assessments are included for all participants but in a sub-study we will consecutively invite participants to also investigate vision and eye functions, brain connectivity and, biomarkers.

PARTICIPANTS PATIENTS All patients present at the Cognitive Post-COVID clinic att the Department of Rehabilitation Medicine at Danderyd University Hospital will have a medical examination. Those patients with cognitive dysfunctions related to a COVID-19 infection will be offered a comprehensive neuropsychological investigation and asked if they are interested in participating in the cohort study.

The first 100 patients are consecutively asked if they also are interested in taking biomarkers. Of these, up to 30 patients, meeting the inclusion criteria for functional Magnetic Resonance Imaging (fMRI) are asked for participation in the a sub-study including an fMRI investigation as well as an optometric and OCT investigation.

NON-SYMPTOMATIC CONTROLS 50 healthy controls who do not suffer from long term symptoms after a COVID-19 infection >3 months from the latest infections or have not had a COVID-19 infection will be investigated for comparison. The same exclusion criteria as for the patients are applied also for the controls. The non-symptomatic controls will undergo neuropsychological examination, examination of visual functions, sampling of biomarkers, as well as fMRI examination and an OCT examination. The controls will be matched with the patients regarding age, gender and length of education.

The patients will be followed-up with questionnaires regarding current symptoms after 1 and 2 years after the neuropsychological investigation.

ELIGIBILITY:
Inclusion Criteria:

• Persons 18 years and older with a history of (> 3 months) verified COVID-19 (PCR / rapid test / antibody) or an infection that is most likely a SARS-CoV-2 infection (e.g., a close relative had a verified infection that coincided in time with the patient's illness) and who have persistent problems with cognitive impairment or fatigue affecting the return to previous activities / employment.

Exclusion Criteria:

* Dominant recurrent and / or fluctuating symptoms of infection, circulatory, respiratory or cardiac problems.
* Co-morbidities that may cause cognitive impairment such as neurodegenerative disease, substance abuse, severe mental illness (eg. schizophrenia, mano depressive disorder) or severe depression.
* Not fluent in Swedish, as test and self-reports rely on good mastering of the Swedish language.
* Severe premorbid visual impairment.

Additionally for the fMRI study:

* Not verified SARS-CoV-2 infection with a Polymerase Chain Reaction (PCR) / rapid test / antibody review
* Traumatic brain injury
* Neuropsychiatric disease such as diagnosed ADHD or autism
* Younger than 25 years or older than 55 years (to avoid the risk that the brain is not fully developed or that there is a risk of age-related changes in the brain).
* MRI contraindications (such as metal objects in the body, fear of cramped spaces, pregnancy, body weight over 130 kg), and left-handedness (to increase the likelihood of uniform topological lateralization in the cohort).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with long term (>3 months) cognitive symptoms and fatigue after a SARS-CoV-2 infection and present at the Department of Rehabilitation Medicine at Danderyd University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigability from Wechsler Adult Intelligence Scale (WAIS)-IV Coding Test | baseline
  The subject must fill in the blank spaces with the symbol which is paired to the number for 120 seconds. Cognitive fatigue is assessed by subtracting the number of digits produced in the first 30 seconds from the number of digits produced in the last 30 seconds during the full 120-second period. A non-ascending score (< 0) is considered an indicator of cognitive fatigue. Both the total value in the difference between the production between 0-30 seconds and 91-120 seconds are measured, and a dichotomized variable (non-ascending value) will be used.
Buschke selective reminding test (BSRT) | baseline
  The BSRT measure verbal learning and long-term memory. The subject hears a list of 12 unrelated words and immediately after that have to recall as many of these 12 words as possible. On each subsequent trial, the subject only hears the words that the subject did not recall on the immediately preceding trial. The test proceed in this manner until the subject can correctly recall all 12 words on two consecutive trials, or until 12 trials have been completed. Through assessing the recall of items that are not presented on a given trial, this test is believed to distinguish between retrieval from long-term storage (LTS) and short-term recall (STR). Consistent recalled words (CLTS) are thought to represent executive aspects of the learning process. After the learning phase, the subject is asked to free recall the words after a 30-minute delay. A cued recall and a multiple-choice condition are also included in the test.
Ruff 2&7 | baseline
  Ruff 2 & 7 measures sustained and selective attention as a continuous performance test during 5 minutes. The subject has to identify and cancel the target digits (2 and 7) among distractors; either letters (automatic sustained attention) or numbers (controlled selective attention), in random order. Both accuracy and speed are measured. Higher scores mean better performance. Performance is evaluated according to the test manual.
The Delis-Kaplan Executive Function System (D-KEFS) Color-Word Test | baseline
  Inhibition of over-learned verbal responses. The test has four conditions: 1) naming colors (red, blue or green, 2) reading color words printed in black, 3) naming the color of the color words red, blue or green write in a different color than what is written, which means inhibition of an over-learned function of reading the word; 4) repeatedly switching between naming colors and reading out the printed words as quickly as possible, while at the same time the person needs to keep track of clues that indicate rule change. Contrast scores are used to examine the performance of the more complex tasks 3 and 4 and the basic tasks 1 and 2. The faster the time, the better
Fatigability on e-prime vigilance task in the fMRI scanner | baseline
  The participants are instructed to push a button as quick as they can when a set of four zeroes appears in a red rectangle and do nothing if other numbers appear. After each response visual feedback of the reaction time is displayed. If the participant reacts at a false stimulus or if the response time of more than 1 sec. the feedback "false answer" or "no answer" is displayed respectively. The stimuli are presented at random intervals.
Task-based fMRI | baseline
  Cerebral perfusion changes during reaction time paradigm.
Resting-state fMRI | baseline
  Changes in functional connectivity after performance of a reaction time paradigm.
Developmental Eye Movement Test | baseline
  Saccadic eye movements are assessed with the Developmental Eye Movement Test. In the first step, the subject read 40 one-digit numbers arranged in two columns. Time duration and reading errors are measured. This is repeated with a new set of numbers where the subject read 80 numbers distributed over 16 horizontal lines. There are 5 irregularly spaced numbers per line, intended to mimic the way the eyes make saccadic movements during reading. For at ratio the total time duration for reading numbers horizontally is divided by the total time for reading numbers vertically.
Visual Motion Sensitivity | baseline
  Sensitivity to movement in the environment was assessed according to the Visual Motion Sensitivity Clinical Test Protocol. The subject is asked to stand and gaze straight ahead at a fixation mark on the wall at eye level at 4 m distance. An Opto Kinetic Nystagmus drum is held at 25 cm from the face. The drum is rotated at slow-medium velocity while the subject is asked to grade symptoms on a scale of 0-10, where zero means no bother at all and 10 a strong effect of nauseous or somatic or visual sensation.
Biomarkers | baseline
  S100B, Astrocyte-derived Extracellular Vesicles (EV) and High Mobility Group Box 1 (Hmbg1). Exploratory targeted analyses using panels of cytokines & chemokines and neuroinflammation will also be used.
Symptom questionnaire | baseline and 1 year and 2 years after the neuropsychological assessment
  The subject rates 32 different cognitive, emotional and physical symptoms where 0 represents have not had this symptom at all, 1 = have had the symptom but is not a problem anymore, 2 = is still a small problem, 3 = is a moderate problem, and 4 = a severe problem. A maximum score is 128 points.
Multidimensional Fatigue Inventory-20 | baseline and 1 year and 2 years after the neuropsychological assessment
  The MFI-20 consists of five scales, based on different modes of expressing fatigue. Each scale contains four items for which the subject indicates on a seven-point scale to what extent the statement applies best. 'General fatigue' includes general statements concerning a person's functioning. 'Physical fatigue' refers to the physical sensation related to the feeling of tiredness. 'Reduced activities' measures reduction in activities and 'Reduced motivation' lack of motivation. 'Mental fatigue' measures cognitive symptoms related to fatigue. Some sentences are inverted and need to be rescored. On each scales the higher values the higher fatigue.
The Montreal Cognitive Assessment (MoCA) | baseline and 1 year and 2 years after the neuropsychological assessment
  A rapid screening test consisting of seven different domains including 1) visuospatial/executive functions, 2) naming, 3) memory, 4) attention, 5) language, 6) abstraction, and 7) orientation. The total score is 30 points +1 point adjustment for low education); normal functioning is considered from score of 26 and above.

SECONDARY OUTCOMES:
Visual Analog Scale of Fatigue | baseline
  Measurement of self-rated current fatigue level. Ranges from 0 (corresponding to no fatigue) to 10 (corresponding to the worst possible fatigue)
D-KEFS Word Fluency Test | baseline
  The test measures expressive language skills, initiative and working memory and consists of three different conditions: verbal phonological flow (1) where the test person for 60 seconds produces as many unique words as possible that begins with a given letter., category flow (2) where the test person for 60 seconds per category produce as many unique words as possible in two given semantic categories and category change (3) where the test person in 60 seconds produce so many unique words and switch between two specified semantic categories every other time. The more words, the better the performance.
WAIS-IV Digit Span | baseline
  The test person must repeat numbers that the test leader reads out the leader reads out. The number of digits is increased by one unit every two times). The test person repeats the numbers in the same order (forward repetition) or reverse order (backward repetition). Forward repetition measures auditory attention span and short-term memory, while backward repetition measures auditory working memory. Both the total number of digits, forward, backward, and the difference between forward and backward repetition will be measured
Convergence Insufficiency Symptom Survey (CISS) | baseline
  Measures symptoms while reading and near activities and intended for symptom assessment in the presence of convergence insufficiency. It includes 15 questions on symptoms and the patient is asked to grade how frequently each symptom occurs: Never (0), Infrequently (1), Sometimes (2), Fairly often (3), or Always (4). A score of 21 is considered useful as a cut-off.
Brain Injury Vision Symptom Survey measuring general vision-related symptoms (BIVSS) | baseline
  BIVSS is originally intended for visual symptom assessment in patients with mild to moderate brain injury. BIVSS includes 28 questions covering seven areas of symptoms: visual clarity/acuity, visual comfort, double vision, photosensitivity, dry eyes, depth perception, visual field, and reading. BIVSS is administered as an interview and for each question the patient is asked to grade how often the symptom occur: Never (0), Seldom (1), Occasionally (2), Frequently (3), or Always (4). A cut-off score of 31 is considered useful for symptom screening.
Rey-Complex Figure Test (RCFT) | baseline
  The RCFT is a visual learning and memory test that also measures other cognitive dimensions, including visuospatial construction skills, fine motor coordination, and planning. The test consists of four subtests: 1) copying, when the subject without time pressure, the time is recorded, is allowed to watch the figure and at the same time depict it without rotating or turning the figure. Immediately afterwards the template is withdrawn, and the subject has to 2) draw the figure again from memory (immediate reproduction). 3) After about 30 minutes (in between, other tests are carried out), the subject must again draw the figure from memory (delayed reproduction), and finally the subject has to 4) select from a booklet possible components from the figure (recognition).
D-KEFS Trail Making Test | baseline
  The TMT measure visual perceptual function, attention, cognitive flexibility, processing speed, and motor speed. The test distinguish whether any weaknesses are due to deficits in underlying skills measured with the subtests 1-3 and 5 (visual scanning, letter or number sequencing or motor speed) or in cognitive flexibility (subtest 4), which is the main measure of the test. The subject is tasked with drawing lines between circles with either letters or numbers or nothing inside. The test subject is asked to complete the tasks as quickly and correctly as possible. The time to perform is measured. The lower score the better the result.
Optical coherence tomography (OCT) | baseline
  Detection of retinal hemorrhages or abnormal retinal layer thickness.

OTHER OUTCOMES:
Sniffn' sticks | baseline
  The Sniffin' Sticks 12 test (Burghardt®, Wedel, Germany) is a smell identification test that measures the ability to recognize 12 common odors. The test is validated in several European countries and has a age and gender separated norms.
Anatomical MRI | baseline
  Abnormal volumetric analyses of the brain. Detection of microvascular pathology.
Other visual functions | baseline
  The vision examination include visual acuity (Snellen Chart, 4 m), near acuity (near chart), stereo acuity (Lang II test), eye motility, and clinical assessment of fixation, pursuit eye movements, and saccadic eye movements (on cue and self-paced). The patient is instructed to keep the head still during eye movement testing and only move the eyes. One or two pens are used as targets and were presented 60 cm from the eyes of the patients. When testing fixation one target is held at 7 positions for 3-4 seconds: primary position, to the left of the patients, up-left, down-left, right, right-up, and right-down. The patient is instructed to maintain fixation on the target as steadily and carefully as possible.
Brief Resilient Coping Scale | baseline
  A 4-item measure designed to capture tendencies to cope with stress in a highly adaptive manner. Scores are ranging from 4-20. The higher scores the better resilience.
WAIS-IV Matrices | baseline
  Matrices measure logical reasoning, visual ability, perceptual organization ability, and the ability to process multiple streams of information simultaneously. The subject is presented with an image of geometric shapes that together form a logical pattern. The test taker is asked to choose from 5 possible solutions the one that best fits into the pattern depicted. The tasks become progressively more difficult.
WAIS-IV Information | baseline
  Information measures the ability to acquire, remember and retrieve general factual knowledge. The subject is instructed to answer a number of general knowledge questions of progressively more and more difficult nature. The subtest measures crystallized intelligence, and is used as a hold test.
Hospital Anxiety and Depression Scale (HADS) | baseline and 1 year and 2 years after the neuropsychological assessment
  HADS (41) consists of two subscales measuring depression (HADS-D) and anxiety (HADS-A). Both subscales range from 0 to 21, with scores> 10 indicating a high risk of depression and anxiety respectively.
Insomnia Severity Index (ISI) Symptoms of disturbed sleep were assessed with ISI (39), | baseline and 1 year and 2 years after the neuropsychological assessment
  ISI is a comprehensive unidimensional self-report scale measuring insomnia on a 5-point Likert scale. The maximal score is 28. Higher values reflect more symptoms and a cut-off score of 10 is optimal in balancing specificity and sensitivity.
The RAND 36-Item Health Survey | baseline and 1 year and 2 years after the neuropsychological assessment
  The RAND 36-Item Health Survey includes eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Borg, Professor, Study Director — Karolinska Institutet; Marika C Möller, PhD, Principal Investigator — Department of Rehabilitation Medicine, Danderyd University Hospital
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsampasian V, Elghazaly H, Chattopadhyay R, Debski M, Naing TKP, Garg P, Clark A, Ntatsaki E, Vassiliou VS. Risk Factors Associated With Post-COVID-19 Condition: A Systematic Review and Meta-analysis. JAMA Intern Med. 2023 Jun 1;183(6):566-580. doi: 10.1001/jamainternmed.2023.0750. PMID 36951832
- [Background] Al-Aly Z, Bowe B, Xie Y. Long COVID after breakthrough SARS-CoV-2 infection. Nat Med. 2022 Jul;28(7):1461-1467. doi: 10.1038/s41591-022-01840-0. Epub 2022 May 25. PMID 35614233
- [Background] Graham EL, Clark JR, Orban ZS, Lim PH, Szymanski AL, Taylor C, DiBiase RM, Jia DT, Balabanov R, Ho SU, Batra A, Liotta EM, Koralnik IJ. Persistent neurologic symptoms and cognitive dysfunction in non-hospitalized Covid-19 "long haulers". Ann Clin Transl Neurol. 2021 May;8(5):1073-1085. doi: 10.1002/acn3.51350. Epub 2021 Mar 30. PMID 33755344
- [Background] Premraj L, Kannapadi NV, Briggs J, Seal SM, Battaglini D, Fanning J, Suen J, Robba C, Fraser J, Cho SM. Mid and long-term neurological and neuropsychiatric manifestations of post-COVID-19 syndrome: A meta-analysis. J Neurol Sci. 2022 Mar 15;434:120162. doi: 10.1016/j.jns.2022.120162. Epub 2022 Jan 29. PMID 35121209
- [Background] Ceban F, Ling S, Lui LMW, Lee Y, Gill H, Teopiz KM, Rodrigues NB, Subramaniapillai M, Di Vincenzo JD, Cao B, Lin K, Mansur RB, Ho RC, Rosenblat JD, Miskowiak KW, Vinberg M, Maletic V, McIntyre RS. Fatigue and cognitive impairment in Post-COVID-19 Syndrome: A systematic review and meta-analysis. Brain Behav Immun. 2022 Mar;101:93-135. doi: 10.1016/j.bbi.2021.12.020. Epub 2021 Dec 29. PMID 34973396
- [Background] Klironomos S, Tzortzakakis A, Kits A, Ohberg C, Kollia E, Ahoromazdae A, Almqvist H, Aspelin A, Martin H, Ouellette R, Al-Saadi J, Hasselberg M, Haghgou M, Pedersen M, Petersson S, Finnsson J, Lundberg J, Falk Delgado A, Granberg T. Nervous System Involvement in Coronavirus Disease 2019: Results from a Retrospective Consecutive Neuroimaging Cohort. Radiology. 2020 Dec;297(3):E324-E334. doi: 10.1148/radiol.2020202791. Epub 2020 Jul 30. PMID 32729812
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Background] Heslin KP, Haruna A, George RA, Chen S, Nobel I, Anderson KB, Faraone SV, Zhang-James Y. Association Between ADHD and COVID-19 Infection and Clinical Outcomes: A Retrospective Cohort Study From Electronic Medical Records. J Atten Disord. 2023 Jan;27(2):169-181. doi: 10.1177/10870547221129305. Epub 2022 Oct 20. PMID 36264064
- [Background] Dobryakova E, DeLuca J, Genova HM, Wylie GR. Neural correlates of cognitive fatigue: cortico-striatal circuitry and effort-reward imbalance. J Int Neuropsychol Soc. 2013 Sep;19(8):849-53. doi: 10.1017/S1355617713000684. Epub 2013 Jul 10. PMID 23842042
- [Background] Nordin LE, Moller MC, Julin P, Bartfai A, Hashim F, Li TQ. Post mTBI fatigue is associated with abnormal brain functional connectivity. Sci Rep. 2016 Feb 16;6:21183. doi: 10.1038/srep21183. PMID 26878885
- [Background] Aceti A, Margarucci LM, Scaramucci E, Orsini M, Salerno G, Di Sante G, Gianfranceschi G, Di Liddo R, Valeriani F, Ria F, Simmaco M, Parnigotto PP, Vitali M, Romano Spica V, Michetti F. Serum S100B protein as a marker of severity in Covid-19 patients. Sci Rep. 2020 Oct 29;10(1):18665. doi: 10.1038/s41598-020-75618-0. PMID 33122776
- [Background] Cantor F. Central and peripheral fatigue: exemplified by multiple sclerosis and myasthenia gravis. PM R. 2010 May;2(5):399-405. doi: 10.1016/j.pmrj.2010.04.012. PMID 20656621
- [Background] Tahyra ASC, Calado RT, Almeida F. The Role of Extracellular Vesicles in COVID-19 Pathology. Cells. 2022 Aug 11;11(16):2496. doi: 10.3390/cells11162496. PMID 36010572
- [Background] Wallensten J, Nager A, Asberg M, Borg K, Beser A, Wilczek A, Mobarrez F. Leakage of astrocyte-derived extracellular vesicles in stress-induced exhaustion disorder: a cross-sectional study. Sci Rep. 2021 Jan 21;11(1):2009. doi: 10.1038/s41598-021-81453-8. PMID 33479350
- [Background] Kanberg N, Ashton NJ, Andersson LM, Yilmaz A, Lindh M, Nilsson S, Price RW, Blennow K, Zetterberg H, Gisslen M. Neurochemical evidence of astrocytic and neuronal injury commonly found in COVID-19. Neurology. 2020 Sep 22;95(12):e1754-e1759. doi: 10.1212/WNL.0000000000010111. Epub 2020 Jun 16. PMID 32546655
- [Background] Bruck E, Lasselin J; HICUS study group; Andersson U, Sackey PV, Olofsson PS. Prolonged elevation of plasma HMGB1 is associated with cognitive impairment in intensive care unit survivors. Intensive Care Med. 2020 Apr;46(4):811-812. doi: 10.1007/s00134-020-05941-7. Epub 2020 Feb 26. No abstract available. PMID 32103282
- [Background] Okuma Y, Wake H, Teshigawara K, Takahashi Y, Hishikawa T, Yasuhara T, Mori S, Takahashi HK, Date I, Nishibori M. Anti-High Mobility Group Box 1 Antibody Therapy May Prevent Cognitive Dysfunction After Traumatic Brain Injury. World Neurosurg. 2019 Feb;122:e864-e871. doi: 10.1016/j.wneu.2018.10.164. Epub 2018 Nov 2. PMID 30391757
- [Background] Ariza M, Cano N, Segura B, Adan A, Bargallo N, Caldu X, Campabadal A, Jurado MA, Mataro M, Pueyo R, Sala-Llonch R, Barrue C, Bejar J, Cortes CU; NAUTILUS-Project Collaborative Group; Junque C, Garolera M. Neuropsychological impairment in post-COVID condition individuals with and without cognitive complaints. Front Aging Neurosci. 2022 Oct 20;14:1029842. doi: 10.3389/fnagi.2022.1029842. eCollection 2022. PMID 36337708
- [Background] Kelly KM, Anghinah R, Kullmann A, Ashmore RC, Synowiec AS, Gibson LC, Manfrinati L, de Araujo A, Spera RR, Brucki SMD, Tuma RL, Braverman A, Kiderman A. Oculomotor, vestibular, reaction time, and cognitive tests as objective measures of neural deficits in patients post COVID-19 infection. Front Neurol. 2022 Sep 12;13:919596. doi: 10.3389/fneur.2022.919596. eCollection 2022. PMID 36188407
- [Background] Marinho PM, Marcos AAA, Romano AC, Nascimento H, Belfort R Jr. Retinal findings in patients with COVID-19. Lancet. 2020 May 23;395(10237):1610. doi: 10.1016/S0140-6736(20)31014-X. Epub 2020 May 12. No abstract available. PMID 32405105
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Sinclair VG, Wallston KA. The development and psychometric evaluation of the Brief Resilient Coping Scale. Assessment. 2004 Mar;11(1):94-101. doi: 10.1177/1073191103258144. PMID 14994958
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Wechsler D. WAIS-IV technical and interpretive manual. San Antonio, Tex.: Psychological Corporation: Pearson; 2008.
- [Background] Delis DC, Kaplan E, Kramer JH. D-KEFS. Examiner´s manual. San Antonio: The Psychological Corporation, a Harcourt Assessment Company; 2001.
- [Background] Kobal G, Hummel T, Sekinger B, Barz S, Roscher S, Wolf S. "Sniffin' sticks": screening of olfactory performance. Rhinology. 1996 Dec;34(4):222-6. PMID 9050101
- [Background] Buschke H. Selective reminding for analysis of memory and learning. Journal of Verbal Learning & Verbal Behavior. 1973;12(5):543-50.
- [Background] Meyers JE, Meyers KR. Rey Complex Figure Test and Recognition Trial Professional Manual. Odessa: Psychological Assessment Resources, Inc. ; 1995.
- [Background] Ruff RM, Allen CC. Ruff 2 & 7 Selective Attention Test. Lutz: Psychological Assessment Resources, Inc.; 1996.
- [Background] Garzia RP, Richman JE, Nicholson SB, Gaines CS. A new visual-verbal saccade test: the development eye movement test (DEM). J Am Optom Assoc. 1990 Feb;61(2):124-35. PMID 2313029
- [Background] Moller MC, Nordin LE, Bartfai A, Julin P, Li TQ. Fatigue and Cognitive Fatigability in Mild Traumatic Brain Injury are Correlated with Altered Neural Activity during Vigilance Test Performance. Front Neurol. 2017 Sep 21;8:496. doi: 10.3389/fneur.2017.00496. eCollection 2017. PMID 28983280
- [Background] Rouse MW, Borsting EJ, Mitchell GL, Scheiman M, Cotter SA, Cooper J, Kulp MT, London R, Wensveen J; Convergence Insufficiency Treatment Trial Group. Validity and reliability of the revised convergence insufficiency symptom survey in adults. Ophthalmic Physiol Opt. 2004 Sep;24(5):384-90. doi: 10.1111/j.1475-1313.2004.00202.x. PMID 15315652
- [Background] Laukkanen H, Scheiman M, Hayes JR. Brain Injury Vision Symptom Survey (BIVSS) Questionnaire. Optom Vis Sci. 2017 Jan;94(1):43-50. doi: 10.1097/OPX.0000000000000940. PMID 28027193
- [Background] Lim J, Wu WC, Wang J, Detre JA, Dinges DF, Rao H. Imaging brain fatigue from sustained mental workload: an ASL perfusion study of the time-on-task effect. Neuroimage. 2010 Feb 15;49(4):3426-35. doi: 10.1016/j.neuroimage.2009.11.020. Epub 2009 Nov 24. PMID 19925871